CLINICAL TRIAL: NCT06287476
Title: Alveolar-capillary Reserve After Exercise in COPD
Brief Title: Alveolar-capillary Reserve After Exercise in Chronic Obstructive Pulmonary Disease (COPD) (COP-DTPA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Ronan Berg, MD, DMSc, Associate Professor, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H-23043870
Record Dates: First submitted 2024-02-12; First posted 2024-03-01 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2024-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Alveolar-capillary membrane integrity; Lung tissue mass; Cardiac Output; DLCO/DLNO
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): This arm consist of only healthy participants (age (+/- 3 years) and sex matched to the COPD group), which will undergo three study visits
  Interventions: Other: Acute exercise bout on visit 2 and 3
- COPD group (Experimental): This arm consist of only COPD patients, which will undergo three study visits
  Interventions: Other: Acute exercise bout on visit 2 and 3

INTERVENTIONS:
Other: Acute exercise bout on visit 2 and 3 — 1) a 5-minute warm-up, 2) 4 minutes at 60% of the maximal workload (determined on Study Day 1), 3) 2 minutes active break at 15 watt, 4) 4 minutes at maximal workload.

SUMMARY:
It is unknown whether individuals with COPD exhibit abnormal alveolar-capillary breaching during exercise, and whether this contributes to exertional dyspnoea. The aim of this study is to investigate whether individuals with COPD exhibit an abnormal increase in alveolar-capillary breaching during exertion, as indicated by an increase alveolar-capillary permeability with a concomitantly exacerbated increase in lung tissue mass.

DETAILED DESCRIPTION:
It is unknown whether individuals with COPD exhibit abnormal alveolar-capillary breaching during exercise, and whether this contributes to exertional dyspnoea. The aim of this study is to investigate whether individuals with COPD exhibit an abnormal increase in alveolar-capillary breaching during exertion, as indicated by an increase alveolar-capillary permeability with a concomitantly exacerbated increase in lung tissue mass. The study participants include a control group and a group with COPD (GOLD I-III). Participants are undergoing three study days: (1) Measurement of maximal aerobic capacity and lung function test, (2) lung tissue mass and alveolar-capillary permeability is measured at rest and again 2 hours later, immediately after the participant has exercised on a bicycle ergometer and (3) supine cardiac output and pulmonary capillary blood volume will be measured at rest and immediately after exercise.

ELIGIBILITY:
Inclusion criteria - individuals with COPD

* Men and women
* 45-80 years old
* COPD (GOLD stage I to III)
* Resting arterial oxygenation > 90%

Inclusion criteria - healthy controls

* Men and women
* 45-80 years old
* Non-smokers
* Normal lung function
* Same sex, age (± 3 years) as the COPD group

Exclusion criteria - individuals with COPD

* Symptoms of ischemic heart disease
* Known heart failure
* Symptoms of illness, including fever, within 2 weeks prior to the study
* Pregnancy
* • Known renal or liver diseaseActive smoking (within 3 weeks)

Exclusion criteria - healthy controls

* Known chronic lung disease
* Symptoms of ischemic heart disease
* Known heart failure
* Symptoms of illness, including fever, within 2 weeks prior to the study
* Pregnancy
* Known renal or liver disease
* Active smoking (within 3 weeks)

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
Rest-to-exercise pulmonary DTPA clearance change after exercise in COPD vs. controls | Measured at study day 2
  The physiological change from rest to exercise in DTPA clearance

SECONDARY OUTCOMES:
Pulmonary DTPA clearance at rest in COPD vs. controls | Measured at study day 2
  Pulmonary DTPA clearance measured by pulmonary DTPA clearance at rest
Pulmonary DTPA clearance after exercise in COPD vs. controls | Measured at study day 2
  Pulmonary DTPA clearance measured by pulmonary DTPA clearance after exercise
Rest-to-exercise change in lung tissue mass in COPD vs. controls | Measured at study day 2
  The physiological change from rest to exercise in lung tissue mass measured by low-dose CT-scan

OTHER OUTCOMES:
Lung tissue mass at rest in COPD vs. controls | Measured at study day 2
  Lung tissue mass measured at rest by low-dose CT-scan
Lung tissue mass after exercise in COPD vs. controls | Measured at study day 2
  Lung tissue mass measured at exercise by low-dose CT-scan
Rest-to-exercise pulmonary DTPA clearance and lung tissue mass change according to GOLD | Measured at study day 2
  The physiological change from rest to exercise in lung tissue mass measured by low-dose CT-scan and the physiological change from rest to exercise in DTPA clearance according to different GOLD stages
Supine pulmonary capillary blood volume after exercise in COPD vs. controls | Measured at study day 3
  Pulmonary capillary blood volume (VC) after exercise obtained by combined DLCO/NO technique with 5-sec breath-hold
Supine cardiac output after exercise in COPD vs. controls | Measured at study day 3
  Cardiac output measured after exercise by a Finometer device
Supine pulmonary capillary blood volume at rest in COPD vs. controls | Measured at study day 3
  VC at rest obtained by combined DLCO/NO technique with 5-sec breath-hold
Supine cardiac output at rest in COPD vs. controls | Measured at study day 3
  Cardiac output measured at rest by a Finometer device
Supine pulmonary diffusing capacity to nitric oxide (DLNO) after exercise in COPD vs. controls | Measured at study day 3
  DLNO measured after exercise by combined DLCO/NO technique with 5-sec breath-hold
Supine haemoglobin-corrected pulmonary diffusing capacity to carbon monoxide (DLCOc) after exercise in COPD vs. controls | Measured at study day 3
  DLCOc measured after exercise by combined DLCO/NO technique with 5-sec breath-hold
Supine alveolar-capillary membrane diffusing capacity (DM) after exercise in COPD vs. controls | Measured at study day 3
  Membrane diffusion capacity (DM) after exercise obtained by combined DLCO/NO technique with 5-sec breath-hold
Supine pulmonary diffusing capacity to nitric oxide (DLNO) at rest in COPD vs. controls | Measured at study day 3
  DLNO measured at rest by combined DLCO/NO technique with 5-sec breath-hold
Supine haemoglobin-corrected pulmonary diffusing capacity to carbon monoxide (DLCOc) at rest in COPD vs. controls | Measured at study day 3
  DLCOc measured at rest by combined DLCO/NO technique with 5-sec breath-hold
Supine alveolar-capillary membrane diffusing capacity (DM) at rest in COPD vs. controls | Measured at study day 3
  DM after exercise obtained by combined DLCO/NO technique with 5-sec breath-hold

CONTACTS AND LOCATIONS:
Locations (1):
- Center For Physical Activity Research, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No